CLINICAL TRIAL: NCT05343351
Title: The Effect of Out of Plane and In Plane Injection Techniques on Injection Pain and Functionality in Patients With Carpal Tunnel Syndrome Undergoing Ultrasound-Guided Injection: A Randomized, Double-Blind Study
Brief Title: Effect of Out of Plane and In Plane Injection Techniques in Patients With Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Alper mengi, Medical Doctor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25.03.2022/109
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Carpal Tunnel Syndrome; Pain; Carpal Tunnel
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain; Median Neuropathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Out of Plane arm (Experimental): The patient group who was injected using the ultrasound-guided out of plane injection method.
  Interventions: Other: Technique of injection method
- In Plane arm (Experimental): The group of patients who were injected using the ultrasound-guided in-plane injection method.
  Interventions: Other: Technique of injection method

INTERVENTIONS:
Other: Technique of injection method — In 'out of plane group', the ultrasound probe will be placed at the entrance level of the proximal carpal tunnel (scaphoid-pisiform plane), the ulnar edge of the median nerve will be taken to the midpoint of the probe, and then the needle will be inserted from the middle point of the probe with the out of plane method. Then the needle will be advanced towards the ulnar side of the median nerve and the injection content will be given into the tunnel.
  In 'in plane group group', the ultrasound probe will be placed at the proximal carpal tunnel entrance level (scaphoid-pisiform plane), it will be entered at a cross angle between the ulnar artery and the median nerve with the in-plane method, and be advanced under the median nerve, and then the injection content will be given into the carpal tunnel.

SUMMARY:
The aim of this study, using two different injection techniques,

1. To evaluate the patients in terms of the pain they feel during the application of carpal tunnel syndrome (CTS) injection,
2. Evaluation in terms of undesirable effects developing after injection,
3. To evaluate the degree of pain/drowsiness, symptom severity and functionality, and median nerve diameter at the end of the first month after the injection, and to evaluate the relationship of these parameters with the pain felt by the patients during the injection.

DETAILED DESCRIPTION:
Among the evaluated patients, the patients who met the inclusion and exclusion criteria and accepted the carpal tunnel syndrome injection will be randomized into 2 groups using the random numbers table.

One group will be injected using the out-of-plane technique under ultrasound, and the other group will be injected using the in-plane technique. Patients will be evaluated before the treatment, at the 1st hour after the injection and at the end of the 4th week after the injection.

Randomization and injection of the patients will be done by Dr Gül Tuğba Bulut, while the evaluation of the patients and the sonographic evaluation of the median nerve will be done by Dr Alper Mengi.

Age, gender, education level, body mass index, duration of symptoms, dominant hand, injection hand, and carpal tunnel syndrome severity detected in EMG of the patients included in the study will be recorded.

The patients will be questioned about the pain they feel during the injection at the end of the 1st hour after the injection, while the degree of pain/numbness in the wrist and finger, symptom severity and functionality, and median nerve diameter are evaluated at the end of the 4th week before and after the injection.

Patients will be questioned about undesirable effects at the end of the 4th week after the injection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Numbness and tingling in the median nerve innervation area with or without pain
* Worsening of symptoms at night
* Positive Tinel and/or Phalen sign
* Symptom duration longer than 12 weeks
* Electrophysiologically mild or moderate CTS being diagnosed.

Exclusion Criteria:

* Presence of conditions such as cervical radiculopathy, polyneuropathy, brachial plexopathy, thoracic outlet syndrome that may mimic CTS
* Presence of multiple entrapment neuropathy
* Weakness in hand thumb abduction or opposition
* Thenar atrophy
* Presence of wrist corticosteroid and/or local anesthetic injection
* Regular use of medical treatment such as oral corticosteroids or NSAIDs
* Having entered a physical therapy program due to CTS in the last 6 months before the injection
* A history of trauma or arthritis attack at the wrist level
* Previous surgery due to CTS
* Thyroid diseases, diabetes, chronic kidney failure
* Having bifid median nerve, persistent median artery, ganglion cyst, tenosynovitis or tendinitis on wrist USG
* Rheumatological disease (rheumatoid arthritis, ankylosing spondylitis, systemic lupus) erythematosus, vasculitis, systemic sclerosis, dermatomyositis)
* Presence of malignancy
* Pregnant or breastfeeding mothers
* Infection or skin lesion at the injection site
* Use of wrist splints in the last 4 weeks
* Allergy to corticosteroids or local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Assessment of pain during injection | 1 hour
  Patients will be asked to rate the average level of pain they feel during the injection as absent, mild, moderate, severe, and unbearable.
Pain/Numbness Evaluation | 3 days
  The severity of pain and numbness of the patients will be questioned by visual analog scale (VAS). A horizontal straight line 10 cm long will be used in the VAS assessment. The patient will be told that a value of 0 represents no pain and numbness, and a value of 10 represents the most severe pain and numbness he has ever felt. In each evaluation, the average of the day and night pain/numbness severity over the last 3 days will be questioned.
Evaluation of symptom severity and functionality | 3 days
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) with Turkish validity and reliability will be used to evaluate the symptom severity and functionality of the patients. BCTQ is a self-filled questionnaire consisting of two parts: symptom severity scale (SSS) and functional status scale (FSS). Each item in both sections has five different answers that score between 1 and 5. The mean score is obtained by dividing the total score by the number of questions and ranges from 1 to 5, with a higher score indicating severe symptom. Average scores are calculated separately for symptom severity and functional status.
Evaluation of undesirable effects | 1 day
  At the controls at the end of the 4th week after the injection, the patients had skin discoloration or fat atrophy, steroid exacerbation (transient pain that started at the 24th hour after the injection and lasted an average of 2-5 days after the injection), superficial infection and median nerve irritation (from the injection). Finger numbness or weakness lasting more than 2 weeks after injection, increasing compared to pre-injection) will be evaluated.
Sonographic evaluation of the median nerve | 1 day
  Ultrasonographic evaluation will be performed with an 18-6 MHz superficial linear probe (Esaote MyLab Five LA435 Transducer). Fixed frequency and depth settings will be used for all measurements. During the examination, patients will be performed in a sitting position facing the clinician, with the elbow in 90° flexion, the forearm supinated, and the fingers in the semi-flexion position. The examination will begin by seeing the median nerve in the axial plane at the wrist localization, and the cross-sectional area of the median nerve (MSCA) will be measured with the probe at the level of the psiform and scaphoid bone. In the measurements, the hyperechoic sheath will be excluded from the drawing and the manual trace method available in the USG device will be used. Square millimeter (mm2) unit will be used for area values in all measurements. All measurements will be made in triplicate and the average of the three measurements will be taken.
Descriptive information | 1 day
  Age, gender, education level, body mass index, duration of symptoms, dominant hand, injection hand, and CTS severity detected in EMG of the patients included in the study will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No